CLINICAL TRIAL: NCT00839982
Title: Study of Oral Clofarabine Plus Low-dose Cytarabine in Previously Treated AML and High-Risk MDS Patients at Least 60 Years of Age
Brief Title: Clofarabine and Cytarabine in Treating Older Patients With AML or High-Risk MDS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2302.00; NCI-2010-00039 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH)
Record Dates: First submitted 2009-02-07; First posted 2009-02-10 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Myelodysplastic Syndrome With Isolated Del(5q); Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Chromosome 5q Deletion Syndrome; Leukemia, Myeloid, Acute | interventions — Clofarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemotherapy) (Experimental): Patients receive clofarabine PO QD on days 1-5 and low-dose cytarabine SC BID on days 1-10 or SC QD on days 1-14. Treatment repeats every 21-28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: clofarabine; Drug: cytarabine

INTERVENTIONS:
Drug: clofarabine — Given PO
  Other Names: CAFdA; Clofarex; Clolar
Drug: cytarabine — Given SC
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside

SUMMARY:
This phase I/II trial studied the side effects and best dose of clofarabine when given together with cytarabine and to see how well they work in treating older patients with acute myeloid leukemia (AML) or high-risk myelodysplastic syndromes (MDS) that have relapsed or not responded to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) of oral clofarabine when given with LDAC (cytarabine) in patients age >= 60 with previously treated AML or high risk MDS.

SECONDARY OBJECTIVES:

I. To determine the response rate, disease-free survival (DFS), and overall survival (OS) after therapy with oral clofarabine and LDAC for previously treated AML or high-risk MDS.

OUTLINE: This is a phase I, dose-escalation study of clofarabine followed by a phase II study.

Patients receive clofarabine orally (PO) once daily (QD) on days 1-5 and low-dose cytarabine subcutaneously (SC) twice daily (BID) on days 1-10 or SC QD on days 1-14. Treatment repeats every 21-28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1st relapse or refractory AML; or patients with high risk MDS (10-19% blasts) who have received previous therapy 1st remission must have been < 1 year
* Must not have received previous ara-C (cytarabine) or clofarabine
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Not candidates for standard 7 + 3 regimen (Ara-C and an anthracycline), high dose Ara-C, or hematopoietic stem-cell transplantation
* Serum creatinine =< 1.0 mg/dL; if serum creatinine > 1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be > 50 L/min/1.73 m^2 as calculated by the Modification of Diet in Renal Disease equation
* Serum bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment
* Male and female patients should use an effective contraceptive method during the study and for a minimum of 6 months after study treatment

Exclusion Criteria:

* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol
* Patients with acute promyelocytic leukemia (APL)
* Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before study entry with the exception of hydroxyurea; the patient must have recovered from all acute toxicities from any previous therapy
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Pregnant or lactating patients
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results
* Have had a diagnosis of another malignancy, unless the patient has been disease free for at least 3 years following the completion of curative intent therapy including the following:

  * Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed.
  * Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated, or a radical prostatectomy or definitive radiotherapy has been performed
* Have currently active gastrointestinal disease, or prior surgery that may affect the ability of the patient to absorb oral clofarabine

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pagel, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Patients receive clofarabine 10mg PO QD on days 1-5 and low-dose cytarabine SC BID on days 1-10 or SC QD on days 1-14. Treatment repeats every 21-28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  clofarabine: Given PO
  cytarabine: Given SC
- Dose Level 2: Patients receive clofarabine 20mg PO QD on days 1-5 and low-dose cytarabine SC BID on days 1-10 or SC QD on days 1-14. Treatment repeats every 21-28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  clofarabine: Given PO
  cytarabine: Given SC
- Dose Level 3: Patients receive clofarabine 25mg PO QD on days 1-5 and low-dose cytarabine SC BID on days 1-10 or SC QD on days 1-14. Treatment repeats every 21-28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  clofarabine: Given PO
  cytarabine: Given SC
- Dose Level 4: Patients receive clofarabine 30mg PO QD on days 1-5 and low-dose cytarabine SC BID on days 1-10 or SC QD on days 1-14. Treatment repeats every 21-28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  clofarabine: Given PO
  cytarabine: Given SC
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Started | 4 | 26 | 2 | 3
Completed | 4 | 26 | 2 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 32
Age, Continuous [Median (Full Range); unit: years] | 72 [62 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicity
Description: Dose limiting toxicity (DLT) consists of grade 3-4 non-hematologic toxicity at least possibly related to study drug. Exceptions include neutropenic fever; drug-related fever; alopecia; anorexia; inadequately treated nausea, vomiting and/or diarrhea; and grade 3/4 increase in ALT, AST, or bilirubin recovering to < grade 2 by 7 days. Prolonged grade 2 myelosuppression lasting longer than 49 days in patients who don't proceed to additional cytotoxic therapy is considered a DLT. The MTD or recommended phase II dose is the highest dose level at which no more than 1 patient out of 6 experiences DLT.
Time Frame: Outcomes by day 30
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1: Patients receive clofarabine 10 mg PO QD on days 1-5 and low-dose cytarabine SC BID on days 1-10 or SC QD on days 1-14. Treatment repeats every 21-28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  clofarabine: Given PO
  cytarabine: Given SC
- Dose Level 2: Patients receive clofarabine 20 mg PO QD on days 1-5 and low-dose cytarabine SC BID on days 1-10 or SC QD on days 1-14. Treatment repeats every 21-28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  clofarabine: Given PO
  cytarabine: Given SC
- Dose Level 3: Patients receive clofarabine 25 mg PO QD on days 1-5 and low-dose cytarabine SC BID on days 1-10 or SC QD on days 1-14. Treatment repeats every 21-28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  clofarabine: Given PO
  cytarabine: Given SC
- Dose Level 4: Patients receive clofarabine 30 mg PO QD on days 1-5 and low-dose cytarabine SC BID on days 1-10 or SC QD on days 1-14. Treatment repeats every 21-28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  clofarabine: Given PO
  cytarabine: Given SC
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 4 | 26 | 2 | 3
Participants | 0 | 4 | 2 | 2
Statistical Analysis 1: Comparison: Dose Level 1; Test type: Superiority; p = 0.03, Chi-squared — Hypothesis: achieving CR provides an overall longer survival

2. Primary Outcome: Maximum Tolerated Dose
Description: We identified 20 mg/d for 5 d as the maximum tolerated dose (MTD) of oral clofarabine.
Time Frame: up to 5 years
Measure: Number; unit: mg/day
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 35
mg/day | 20

3. Secondary Outcome: Treatment Response
Description: CR = no evidence of leukemia with complete blood count recovery (ANC >1,000 and PLTS >100k) CRi = no evidence of leukemia but with incomplete blood count recovery
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 4 | 26 | 2 | 3
Participants
  CR | 1 | 10 | 1 | 0
  CRi | 0 | 1 | 0 | 0
  No CR | 3 | 15 | 1 | 3

4. Secondary Outcome: Disease Free Survival
Description: Median disease-free survival
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: median months
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 35
median months | 7.4 [0 to 11]

5. Secondary Outcome: Overall Survival
Description: Median overall survival
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: median months
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 35
median months | 6.8 [1 to 47]

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse events were not reported by dose level.
Groups:
- Treatment (Chemotherapy): Patients receive clofarabine PO QD on days 1-5 and low-dose cytarabine SC BID on days 1-10 or SC QD on days 1-14. Treatment repeats every 21-28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  clofarabine: Given PO cytarabine: Given SC
Arm/Group | Treatment (Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 5/35
Serious Adverse Events (participants affected / at risk) | 24/35
Other Adverse Events (participants affected / at risk) | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy) (N=35)
Infections (Infections and infestations) | 24 (24)
Febrile neutropenia (General disorders) | 8 (8)
Septic Shock (General disorders) | 5 (5)
Bacteraemia (Infections and infestations) | 10 (10)
Bacterial infection other than blood (Infections and infestations) | 7 (7)
Fungal infection (Infections and infestations) | 2 (2)
Arrhythmia (Cardiac disorders) | 3 (3)
Altered Mental Status (Nervous system disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1)
Syncope (General disorders) | 1 (1)
Stroke (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes